CLINICAL TRIAL: NCT00968201
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Chronic Asthma Study Comparing Montelukast With Placebo in 2- to 5-Year-Old Patients
Brief Title: Chronic Asthma Study in 2- to 5-Year-Old Patients (MK0476-072 )
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-072; 2009_651
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Montelukast
  Interventions: Drug: montelukast sodium
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast sodium — one chewable 4-mg montelukast tablet, once daily at bedtime for 12 weeks
  Arms: 1
Drug: Comparator: Placebo — one chewable placebo tablet, once daily at bedtime for 12 weeks
  Arms: 2

SUMMARY:
A study in 2-5 year old children to evaluate the safety and tolerability of montelukast and placebo administered once daily at bed time.

ELIGIBILITY:
Inclusion Criteria:

* Patient has history of physician diagnosed asthma
* Patient is in otherwise good stable health
* Patient is able to chew a tablet

Exclusion Criteria:

* Patient is hospitalized
* Patient and/or parent of guardian intends to move or vacation away from home during the course of the study
* Patient had any major surgical procedure within 4 weeks before the study
* Patient had active sinus disease within 3 weeks before the study
* Patient had required intubation for asthma in the past
* Patient required a visit to the emergency room due to an asthma exacerbation, or has been hospitalized for asthma with in 1 month prior to the study
* Patient had used inhaled, nebulized, intramuscular, or intravenous steroids with in 1 month before study

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 689 (Actual)
Dates: Start 1997-12; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Knorr B, Franchi LM, Bisgaard H, Vermeulen JH, LeSouef P, Santanello N, Michele TM, Reiss TF, Nguyen HH, Bratton DL. Montelukast, a leukotriene receptor antagonist, for the treatment of persistent asthma in children aged 2 to 5 years. Pediatrics. 2001 Sep;108(3):E48. doi: 10.1542/peds.108.3.e48. PMID 11533366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Base Study: 93 sites in the United States (US) and other countries in Africa, Australia, Europe, North America, and South America. Therapy period: Dec-1997 to Mar-1999.
  Extension Study: 75 sites in the US and other countries in Africa, Australia, Europe, North America, and South America. Therapy period: Mar-1998 to Mar-2001.
Pre-assignment Details: Base Study: Patients who required excluded medication and those who did not meet a minimum predefined level of asthma symptoms and β-agonist use during run-in (Period I) were excluded from randomization (Period II).
  Extension Study (Period III): Patients who did not complete Visit 9 of Base Study were not eligible for the optional Extension.
Groups:
- Placebo: Montelukast matching-image placebo chewable tablet orally once daily at bedtime for 12 weeks.
- Usual Care: "Usual care," defined as inhaled/nebulized cromolyn or inhaled/nebulized corticosteroids according to the usual clinical practice of the investigator, for up to 2.8 years. Some patients receiving placebo in Period II were switched to usual care in the Extension Study, and some
  patients receiving montelukast in Period II were switched to usual care in the Extension Study.
  Patients already using corticosteroids during Period I and II continued on the same medication and dose throughout Period II. Their dose was not increased if they were allocated to the "usual care" treatment group in Period III.
- Montelukast: Base Study - Montelukast 4 mg chewable tablet orally once daily at bedtime for 12 weeks.
  Extension Study - Montelukast 4 mg chewable tablet orally once daily at bedtime for up to 2.8 years. Some patients receiving placebo in Period II were switched to montelukast in the Extension Study, and some patients receiving montelukast in Period II continued on montelukast in the Extension Study. One hundred sixty-seven patients were switched to the 5 mg chewable tablet at
  their first visit after turning 6 years old. The 4 mg and 5 mg chewable tablet data are pooled together.
Period: Base Study - (Period II)
Arm/Group | Placebo | Usual Care | Montelukast
Started | 228 (Includes patients who completed Period I (2-week placebo run-in) and were randomized to placebo.) | 0 | 461 (Includes patients who completed Period I (2-week placebo run-in) and were randomized to montelukast.)
Completed | 202 (Patients completing Period II were eligible to enter the optional Period III) | 0 | 416 (Patients completing Period II were eligible to enter the optional Period III)
Not Completed | 26 | 0 | 45
Not completed — Adverse Event | 8 | 0 | 16
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 7
Not completed — Protocol Violation | 12 | 0 | 12
Not completed — Withdrawal by Subject | 4 | 0 | 8
Not completed — Site Error | 0 | 0 | 1
Period: Extension Study - (Period III)
Arm/Group | Placebo | Usual Care | Montelukast
Started | 0 | 157 (Eligible Patients who completed Period II and entered the optional Extension Study (Period III)) | 364 (Eligible Patients who completed Period II and entered the optional Extension Study (Period III))
Completed | 0 | 33 | 84
Not Completed | 0 | 124 | 280
Not completed — Adverse Event | 0 | 5 | 22
Not completed — Lost to Follow-up | 0 | 7 | 13
Not completed — Protocol Violation | 0 | 17 | 14
Not completed — Withdrawal by Subject | 0 | 20 | 40
Not completed — Patient Relocated | 0 | 1 | 1
Not completed — Noncompliance | 0 | 0 | 3
Not completed — Other | 0 | 0 | 2
Not completed — Study Terminated for Admin Reasons | 0 | 74 | 185

BASELINE CHARACTERISTICS:
Groups:
- Montelukast: Base Study - Montelukast 4 mg chewable tablet orally once daily at bedtime for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast | Total
Number analyzed (Participants) | 228 | 461 | 689
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.62 (1.10) | 3.58 (1.11) | 3.59 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 189 | 286
  Male | 131 | 272 | 403

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAE) Reported by Patients - Base Study
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  With CAEs | 202 | 406
  Without CAEs | 26 | 55

2. Secondary Outcome: Number of Patients With Drug-related CAEs Reported by Patients - Base Study
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
  Drug relationship for 1 patient in the Placebo group should have been listed as definitely not drug related.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  With Drug-Related CAEs | 9 | 19
  Without Drug-Related CAEs | 219 | 442

3. Secondary Outcome: Number of Patients With Serious CAEs Reported by Patients - Base Study
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
  A serious CAE (study drug overdose) prior to randomization in the Placebo group is not included in this number
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  With Serious CAEs | 9 | 17
  Without Serious CAEs | 219 | 444

4. Secondary Outcome: Number of Patients With Serious Drug-related CAEs Reported by Patients - Base Study
Description: Patients who reported serious drug-related CAEs during 12 weeks of treatment
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  With Serious Drug-related CAEs | 0 | 2
  Without Serious Drug-related CAEs | 228 | 459

5. Secondary Outcome: Number of Patients Who Were Discontinued Due to CAEs - Base Study
Description: Patients who were discontinued due to CAEs during 12 weeks of treatment
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  Discontinued Due to CAEs | 7 | 16
  Did Not Discontinue Due to CAEs | 221 | 445

6. Secondary Outcome: Number of Patients Who Were Discontinued Due to Drug-related CAEs - Base Study
Description: Patients who were discontinued due to drug-related CAEs during 12 weeks of treatment
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  Discontinued Due to Drug-related CAEs | 1 | 2
  Did Not Discontinue Due to Drug-related CAEs | 227 | 459

7. Secondary Outcome: Number of Patients Who Were Discontinued Due to Serious CAEs - Base Study
Description: Patients who were discontinued due to serious CAEs during 12 weeks of treatment
Time Frame: 12 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 228 | 461
Participants
  Discontinued Due to Serious CAEs | 2 | 8
  Did Not Discontinue Due to Serious CAEs | 226 | 453

8. Secondary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) - Base Study
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 12 weeks of treatment
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 224 | 451
Participants
  With LAEs | 12 | 16
  Without LAEs | 212 | 435

9. Secondary Outcome: Number of Patients With Drug-related Laboratory Adverse Experiences (LAEs) - Base Study
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) LAEs
Time Frame: 12 weeks of treatment
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 224 | 451
Participants
  With Drug-Related LAEs | 1 | 7
  Without Drug-Related LAEs | 223 | 444

10. Secondary Outcome: Number of Patients Who Were Discontinued Due to LAEs - Base Study
Description: Patients who were discontinued due to LAEs during 12 weeks of treatment
Time Frame: 12 weeks of treatment
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 224 | 451
Participants
  Discontinued Due to LAEs | 1 | 0
  Did Not Discontinue Due to LAEs | 223 | 451

11. Secondary Outcome: Number of Patients Who Were Discontinued Due to Drug-related LAEs - Base Study
Description: Patients who were discontinued due to drug-related LAEs during 12 weeks of treatment
Time Frame: 12 weeks of treatment
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 224 | 451
Participants
  Discontinued Due to Drug-related LAEs | 1 | 0
  Did Not Discontinue Due to Drug-related LAEs | 223 | 451

12. Secondary Outcome: Number of Patients With Clinical Adverse Experiences (CAE) Reported by Patients - Extension
Description: as for outcome 1
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Groups:
- Montelukast: Extension Study - Montelukast 4 mg chewable tablet orally once daily at bedtime for up to 2.8 years. Some patients receiving placebo in Period II were switched to montelukast in the Extension Study, and some patients receiving montelukast in Period II continued on montelukast in the Extension Study. One hundred sixty-seven patients were switched to the 5 mg chewable tablet at their first visit after turning 6 years old. The 4 mg and 5 mg chewable tablet data are pooled together.
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  With CAE | 149 | 353
  Without CAE | 8 | 11

13. Secondary Outcome: Number of Patients With Drug-related CAEs Reported by Patients - Extension
Description: as for outcome 2
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  With Drug-related CAEs | 2 | 14
  Without Drug-related CAEs | 155 | 350

14. Secondary Outcome: Number of Patients With Serious CAEs Reported by Patients - Extension
Description: as for outcome 3
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  With Serious CAEs | 15 | 38
  Without Serious CAEs | 142 | 326

15. Secondary Outcome: Number of Patients With Serious Drug-related CAEs Reported by Patients - Extension
Description: Patients who reported serious drug-related CAEs up to 2.8 years of
  treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  With Serious Drug-related CAEs | 0 | 4
  Without Serious Drug-related CAEs | 157 | 360

16. Secondary Outcome: Number of Patients Who Were Discontinued Due to CAEs - Extension
Description: Patients who were discontinued due to CAEs up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  Discontinued Due to CAEs | 5 | 18
  Did Not Discontinue Due to CAEs | 152 | 346

17. Secondary Outcome: Number of Patients Who Were Discontinued Due to Drug-related CAEs - Extension
Description: Patients who were discontinued due to drug-related CAEs with up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  Discontinued Due to Drug-related CAEs | 0 | 2
  Did Not Discontinue Due to Drug-related CAEs | 157 | 362

18. Secondary Outcome: Number of Patients Who Were Discontinued Due to Serious CAEs - Extension
Description: Patients who were discontinued due to serious CAEs with up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  Discontinued Due to Serious CAEs | 1 | 9
  Did Not Discontinue Due to Serious CAEs | 156 | 355

19. Secondary Outcome: Number of Patients Who Were Discontinued Due to Serious Drug-related CAEs - Extension
Description: Patients who were discontinued due to serious drug-related CAEs with up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 157 | 364
Participants
  Discontinued Due to Serious Drug-related CAEs | 0 | 1
  Not Discontinued Due to Serious Drug-related CAEs | 157 | 363

20. Secondary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) - Extension
Description: as for outcome 8
Time Frame: up to 2.8 years
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  With LAEs | 14 | 42
  Without LAEs | 140 | 315

21. Secondary Outcome: Number of Patients With Drug-related Laboratory Adverse Experiences (LAEs) - Extension
Description: as for outcome 9
Time Frame: up to 2.8 years
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  With Drug-related LAEs | 0 | 7
  Without Drug-related LAEs | 154 | 350

22. Secondary Outcome: Number of Patients With Serious LAEs - Extension
Description: Serious LAEs are any LAEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: up to 2.8 years
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  With Serious LAEs | 0 | 1
  Without Serious LAEs | 154 | 356

23. Secondary Outcome: Number of Patients With Serious Drug-related Laboratory Adverse Experiences (LAEs) - Extension
Description: Patients who reported serious drug-related LAEs up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  With Serious Drug-Related LAEs | 0 | 1
  Without Serious Drug-Related LAEs | 154 | 356

24. Secondary Outcome: Number of Patients Who Were Discontinued Due to LAEs - Extension
Description: Patients who were discontinued due to LAEs up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  Discontinued Due to LAEs | 0 | 4
  Did Not Discontinue Due to LAEs | 154 | 353

25. Secondary Outcome: Number of Patients Who Were Discontinued Due to Drug-related LAEs - Extension
Description: Patients who were discontinued due to drug-related LAEs with up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  Discontinued Due to Drug-related LAEs | 0 | 4
  Did Not Discontinue Due to Drug-related LAEs | 154 | 353

26. Secondary Outcome: Number of Patients Who Were Discontinued Due to Serious LAEs - Extension
Description: Patients who were discontinued due to serious LAEs with up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  Discontinued Due to Serious LAEs | 0 | 1
  Did Not Discontinue Due to Serious LAEs | 154 | 356

27. Secondary Outcome: Number of Patients Who Were Discontinued Due to Serious Drug-related LAEs - Extension
Description: Patients who were discontinued due to serious drug-related LAEs with up to 2.8 years of treatment
Time Frame: up to 2.8 years
Population: All patients who took study medication and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 154 | 357
Participants
  Discontinued Due to Serious Drug-related LAEs | 0 | 1
  Not Discontinued Due to Serious Drug-related LAEs | 154 | 356

ADVERSE EVENTS:
Time Frame: During the 12 week base study (Period II) and 36 month extension study (Period III) and up to and including 14 days after the last dose of study therapy.
Description: Although patient may have had 2 or more clinical adverse experiences, patient is counted only once in a category. The same patient may appear in different categories. Adverse events (AEs) in Period II have 0/0 for Usual Care group because there was no Usual Care group. AEs in Period III have 0/0 for Placebo group because there was no Placebo group.
Arm/Group | Placebo | Usual Care | Montelukast
Serious Adverse Events (participants affected / at risk) | 9/228 | 15/157 | 56/461
Other Adverse Events (participants affected / at risk) | 188/228 | 148/157 | 435/461
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=228) | Usual Care (N=157) | Montelukast (N=461)
Drug Overdose (Period II) (Injury, poisoning and procedural complications) | 3 | 0/0 | 5
Drug Overdose (Period III) (Injury, poisoning and procedural complications) | 0/0 | 0 | 9/364
Infection, Viral (Period III) (Infections and infestations) | 0/0 | 1 | 1/364
Pain, Abdominal (Period III) (General disorders) | 0/0 | 0 | 1/364
Trauma (Period III) (Injury, poisoning and procedural complications) | 0/0 | 0 | 1/364
Tachycardia (Period III) (Injury, poisoning and procedural complications) | 0/0 | 0 | 1/364
Appendicitis (Period III) (Infections and infestations) | 0/0 | 0 | 1/364
Gastroenteritis (Period II) (Gastrointestinal disorders) | 0 | 0/0 | 1
Gastroenteritis, Infectious (Period III) (Infections and infestations) | 0/0 | 0 | 2/364
Gastroesophageal Reflux (Period III) (Gastrointestinal disorders) | 0/0 | 0 | 1/364
Infection, Intra-Abdominal (Period III) (Infections and infestations) | 0/0 | 0 | 1/364
Thirst (Period II) (General disorders) | 0 | 0/0 | 2
Thirst (Period III) (General disorders) | 0/0 | 0 | 2/364
Vomiting (Period III) (Gastrointestinal disorders) | 0/0 | 0 | 1/364
Alkaline Phosphatase Increased (Period III) (Investigations) | 0/0 | 0 | 1/364
Allergy (Period III) (Immune system disorders) | 0/0 | 1 | 0/364
Dehydration (Period II) (Metabolism and nutrition disorders) | 1 | 0/0 | 0
Dehydration (Period III) (Metabolism and nutrition disorders) | 0/0 | 0 | 2/364
Hypokalemia (Period III) (Investigations) | 0/0 | 0 | 1/364
Bipolar Disorder (Period II) (Psychiatric disorders) | 1 | 0/0 | 0
Concussion (Period III) (Injury, poisoning and procedural complications) | 0/0 | 0 | 1/364
Headache (Period III) (Nervous system disorders) | 0/0 | 0 | 1/364
Hyperkinesia (Period III) (Nervous system disorders) | 0/0 | 0 | 1/364
Hypersomnia (Period III) (Nervous system disorders) | 0/0 | 0 | 1/364
Meningitis (Period III) (Infections and infestations) | 0/0 | 0 | 1/364
Seizure Disorder (Period III) (Nervous system disorders) | 0/0 | 0 | 1/364
Somnolence (Period II) (Nervous system disorders) | 0 | 0/0 | 1
Somnolence (Period III) (Nervous system disorders) | 0/0 | 0 | 1/364
Tremor (Period III) (Nervous system disorders) | 0/0 | 0 | 1/364
Apnea (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 1/364
Asthma (Period II) (Respiratory, thoracic and mediastinal disorders) | 5 | 0/0 | 10
Asthma (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 8 | 13/364
Bronchoconstriction (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 2 | 2/364
Hypoxemia (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 1 | 1/364
Infection, Respiratory, Upper (Period II) (Infections and infestations) | 1 | 0/0 | 0
Infection, Respiratory, Upper (Period III) (Infections and infestations) | 0/0 | 0 | 1/364
Infiltrate, Pulmonary (Period II) (Respiratory, thoracic and mediastinal disorders) | 1 | 0/0 | 0
Pneumonia (Period II) (Infections and infestations) | 0 | 0/0 | 1
Pneumonia (Period III) (Infections and infestations) | 0/0 | 3 | 3/364
Pneumonia, Bacterial (Period III) (Infections and infestations) | 0/0 | 1 | 0/364
Pneumonia, Viral (Period III) (Infections and infestations) | 0/0 | 0 | 1/364
Sinusitis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 1 | 0/364
Pallor (Period III) (Skin and subcutaneous tissue disorders) | 0/0 | 0 | 1/364
Infection, Eyelid (Period III) (Infections and infestations) | 0/0 | 0 | 1/364
Mydriasis (Period II) (Eye disorders) | 0 | 0/0 | 1
Anomaly, Urogenital (Period III) (Renal and urinary disorders) | 0/0 | 0 | 1/364
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=228) | Usual Care (N=157) | Montelukast (N=461)
Fever (Period II) (General disorders) | 61 | 0/0 | 125
Fever (Period III) (General disorders) | 0/0 | 60 | 164/364
Infection, Viral (Period III) (Infections and infestations) | 0/0 | 25 | 55/364
Pain, Abdominal (Period II) (General disorders) | 21 | 0/0 | 51
Pain, Abdominal (Period III) (General disorders) | 0/0 | 16 | 46/364
Trauma (Period III) (Injury, poisoning and procedural complications) | 0/0 | 10 | 29/364
Dental Caries (Period III) (Gastrointestinal disorders) | 0/0 | 10 | 12/364
Diarrhea (Period II) (Gastrointestinal disorders) | 17 | 0/0 | 45
Diarrhea (Period III) (Gastrointestinal disorders) | 0/0 | 28 | 58/364
Gastroenteritis (Period III) (Gastrointestinal disorders) | 0/0 | 7 | 21/364
Vomiting (Period II) (Gastrointestinal disorders) | 45 | 0/0 | 75
Vomiting (Period III) (Gastrointestinal disorders) | 0/0 | 28 | 60/364
Allergy (Period III) (Immune system disorders) | 0/0 | 4 | 22/364
Headache (Period II) (Nervous system disorders) | 17 | 0/0 | 35
Headache (Period III) (Nervous system disorders) | 0/0 | 26 | 57/364
Asthma (Period II) (Respiratory, thoracic and mediastinal disorders) | 83 | 0/0 | 130
Asthma (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 96 | 217/364
Bronchitis (Period II) (Respiratory, thoracic and mediastinal disorders) | 18 | 0/0 | 18
Bronchitis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 38 | 58/364
Congestion, Nasal (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 11 | 30/364
Cough (Period II) (Respiratory, thoracic and mediastinal disorders) | 26 | 0/0 | 58
Cough (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 24 | 97/364
Epistaxis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 7 | 25/364
Infection, Respiratory (Period II) (Infections and infestations) | 13 | 0/0 | 19
Infection, Respiratory (Period III) (Infections and infestations) | 0/0 | 16 | 44/364
Infection, Respiratory, Upper (Period II) (Infections and infestations) | 63 | 0/0 | 123
Infection, Respiratory, Upper (Period III) (Infections and infestations) | 0/0 | 81 | 192/364
Influenza (Period III) (Infections and infestations) | 0/0 | 14 | 40/364
Laryngitis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 8 | 22/364
Pharyngitis (Period II) (Respiratory, thoracic and mediastinal disorders) | 35 | 0/0 | 54
Pharyngitis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 50 | 120/364
Pneumonia (Period III) (Infections and infestations) | 0/0 | 7 | 21/364
Rhinitis (Period II) (Respiratory, thoracic and mediastinal disorders) | 14 | 0/0 | 27
Rhinitis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 21 | 45/364
Rhinitis, Allergic (Period II) (Respiratory, thoracic and mediastinal disorders) | 16 | 0/0 | 24
Rhinitis, Allergic (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 13 | 40/364
Rhinorrhea (Period II) (Respiratory, thoracic and mediastinal disorders) | 9 | 0/0 | 35
Rhinorrhea (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 16 | 32/364
Sinus Disorder (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 15 | 16/364
Sinusitis (Period II) (Respiratory, thoracic and mediastinal disorders) | 16 | 0/0 | 33
Sinusitis (Period III) (Respiratory, thoracic and mediastinal disorders) | 0/0 | 43 | 95/364
Tonsillitis (Period II) (Infections and infestations) | 15 | 0/0 | 12
Tonsillitis (Period III) (Infections and infestations) | 0/0 | 28 | 56/364
Rash (Period III) (Skin and subcutaneous tissue disorders) | 0/0 | 8 | 21/364
Urticaria (Period III) (Skin and subcutaneous tissue disorders) | 0/0 | 10 | 32/364
Varicella (Period III) (Skin and subcutaneous tissue disorders) | 0/0 | 20 | 45/364
Conjunctivitis (Period III) (Eye disorders) | 0/0 | 9 | 32/364
Otitis (Period II) (Ear and labyrinth disorders) | 8 | 0/0 | 29
Otitis (Period III) (Ear and labyrinth disorders) | 0 | 33 | 62/364
Otitis Media (Period II) (Ear and labyrinth disorders) | 17 | 0/0 | 36
Otitis Media (Period III) (Ear and labyrinth disorders) | 0/0 | 35 | 84/364
Pain, Ear (Period III) (Ear and labyrinth disorders) | 0/0 | 10 | 25/364

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.